CLINICAL TRIAL: NCT05438810
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of FCN-437c Versus Placebo Combined With Fulvestrant ± Goserelin in Women With HR+ and HER2- Advanced Breast Cancer
Brief Title: This is a Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study Evaluating the Efficacy and Safety of FCN-437c in Combination With Fluvestrant ± Goseraline Versus Placebo Combined With Fulvestrant ± Goserelin in Women With HR+ and HER2- Advanced Breast Cancer.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FCN-437c-III202
Record Dates: First submitted 2022-06-24; First posted 2022-06-30 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Advanced Breast Cancer; Female Breast Cancer
Keywords: HR receptor positive HER2 receptor negative; Combined with flulvestrone ± goseraline
MeSH Terms: interventions — Goserelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCN-437c+Fulvestrant ± Goserelin acetate (Experimental)
  Interventions: Drug: FCN-437c,Fulvestrant,Goserelin acetate
- Placebo+ Fulvestrant ± Goserelin acetate (Placebo Comparator)
  Interventions: Drug: Placebo,Fulvestrant,Goserelin acetate

INTERVENTIONS:
Drug: FCN-437c,Fulvestrant,Goserelin acetate — FCN-437c：available in 25mg and 100mg capsules for oral administration on an empty stomach. 200mg once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment until progressive disease。 Fulvestrant：500mg intramuscular injection on day 1 and day 15 for the first cycle and then on day 1 only for other cycles ； Goserelin acetate：premenopausal /perimenopausal patients should be coadministered with 3.6mg, Subcutaneously at every 28 days until progressive disease。
  Arms: FCN-437c+Fulvestrant ± Goserelin acetate
Drug: Placebo,Fulvestrant,Goserelin acetate — Placebo：available in 25mg and 100mg capsules, and is administered in the same way as FCN-437c。 Fulvestrant：500mg intramuscular injection on day 1 and day 15 for the first cycle and then on day 1 only for other cycles； Goserelin acetate：premenopausal /perimenopausal patients should be coadministered with 3.6mg, Subcutaneously at every 28 days until progressive disease。
  Arms: Placebo+ Fulvestrant ± Goserelin acetate

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase iii clinical study evaluating the efficacy and safety of FCN- 437c in combination with fluvestrant ± goseraline versus placebo in combination with fluvestrant ± goseraline in women with HR+ and HER2- advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following conditions:

1. Female advanced breast cancer patients aged ≥18 years, diagnosed as HR+ HER2-. HR+ positive is defined as：Histological and/or cytological confirmed ER+, PR + or -, defined as immunohistochemistry showing positive nuclear staining of estrogen/progesterone receptor tumor cells≥1%； HER2-negative is defined as：Histological and/or cytological confirmed HER2-， defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+,the ISH test result must be negative。
2. Arbitrary menopausal status.Postmenopausal female is defined as:

   After bilateral oophorectomy ; Age≥60 years Age<60 years and menopause for more than 1 year without chemotherapy and treatment with tamoxifen, toremifene and ovarian function suppression, while blood FSH and estradiol levels meet the postmenopausal range and for postmenopausal patients who are taking tamoxifen or toremifene and who are younger than 60 years old, continuous detection of serum FSH and estradiol levels must meet the postmenopausal range..
3. Previous treatment criteria: Second-line and above patients can be included in the group。
4. Previous treatment criteria: Second-line and above patients can be enrolled. Eastern cooperative oncology group (ECOG) 0-1。
5. According to the RECIST 1.1 criteria, patients must have at least one measurable lesion, or patients with only bone metastases, if no measurable lesions are present, must have at least one bone lesion predominantly lytic.

   Note:If the lesion has received radiotherapy or other locoregional treatment, there must be imaging evidence of disease progression in the lesion after completion of treatment, and the lesion can be considered as a measurable lesion. For patients with no measurable lesion and only one osteolytic lesion, if the lesion was previously treated with radiotherapy, imaging evidence is needed to show the progression of bone lesions after radiotherapy.。
6. Life expectancy is not less than 12 weeks;
7. Adequate bone marrow and organ function:

   1. Absolute neutrophil count (ANC) ≥1.5 x 109/L
   2. Hemoglobin ≥90 g/dL(no red blood cell infusion within 14 days before randomization)
   3. Platelet count ≥90 x 109/L
   4. Total serum bilirubin ≤ 1.5 X upper limit of normal (ULN) , total serum bilirubin≤3 x ULN in patients with Gilbert syndrome;
   5. Aspartate aminotransferase (AST)and alanine aminotransferase (ALT) ≤2.5x ULN; for patients with liver metastases,both AST and ALT ≤5× ULN;
   6. Creatinine <1.5 × ULN or creatinine clearance≥50 mL / min[Ccr = ((140- age) ×body weight (kg)) / (72× Scr (mg / dl)) or Ccr = ((140-age)× body weight (kg)) / (0.818× Scr (umol / L)) Note: Females were calculated ×0.85]
   7. QTcF < 470 ms ；
8. The patient is willing and able to comply with planned visits, treatment plans, laboratory examinations, and other trial procedures。
9. The patient is fully aware of the study and has signed an informed consent form (ICF);
10. For perimenopausal/premenopausal patients only: a high-efficiency contraceptive method with a failure rate of less than 1% per year must be used with a partner throughout the study period and for at least 90 days after discontinuation.

Exclusion Criteria:

Patients who meet any of the following conditions are not allowed to enter this clinical study：

1. The exclusion criteria for prior treatment are as follows

   1. Patients who received prior treatment with any CDK4/6 inhibitors or fulvestrant or everolimus;
   2. Received more than first-line systemic chemotherapy for advanced breast cancer.;
   3. Received endocrine therapy within 2 weeks prior to initial administration;
   4. Received radiotherapy, major surgery, tumor immunotherapy, monoclonal antitumor drug therapy, and other systemic antitumor therapies that the investigator considered would interfere with the efficacy of the investigational drug within 4 weeks prior to initial administration.
2. Patients with visceral crises who are not suitable for endocrine therapy.
3. Inflammatory breast cancer.
4. Presence of clinically uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage or medical intervention (within 2 weeks prior to initial administration).
5. Any other malignancy diagnosed within 3 years prior to participation in this study, except radically treated early stage malignancies (carcinoma in situ or stage I tumors) , such as adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ.
6. Toxic response to prior antineoplastic therapy has not recovered to ≤ grade 1 (NCI-CTCAE version 5.0).
7. Cardiac function and disease conform to one of the following conditions:

   1. During the screening period, 12-lead Electrocardiogram (ECG) measurements are performed at the research center, calculated according to the QTcF formula using the instrument,QTcF interval >470 msec.
   2. Clinically significant arrhythmias, including but not limited to complete left bundle branch block, second-degree atrioventricular block.
   3. Any risk factors that increase QTc prolongation, such as hypokalemia, hereditary long QT syndrome, taking drugs that prolong QTc (mainly including anti-IA, Ic, and class III antiarrhythmic drugs), and drugs that potentially prolong QTc are listed in Appendix 6.
   4. Congestive Heart failure rated grade 2 or higher by the New York Heart Association (NYHA).
8. Dysphagia, or active digestive disease, or major gastrointestinal surgery, or malabsorption syndrome, or other conditions that may impair the absorption of FCN-437C (e.g., ulcerative lesions, uncontrollable nausea, vomiting, diarrhea, malabsorption syndrome and small bowel resection).
9. Known to be allergic to fulvestrant, Goserelin, FCN-437C or any other excipients;
10. Clinically suspected brain metastasis meningeal metastasis or unstable brain parenchymal metastasis, but stable brain metastasis can be enrolled。Stable brain metastasis is defined as: no expansion of the original metastatic lesions and no new lesions are found in the imaging reports at intervals of more than one month;No clinical symptoms, no need for hormone or other dehydrating treatment;
11. Patients with active infection, including those who are positive for hepatitis B surface antigen (HBsAg) and whose HBV DNA quantification is ≥ 1.00 x103 IU/ml；Hepatitis C antibody (anti-HCV) positive patients; patients infected with human immunodeficiency virus (HIV).
12. Any other clinically significant disease or condition (such as uncontrolled diabetes, active or uncontrolled infection, etc.) that the investigator believes may affect protocol compliance or the ICF signature.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-02-18 (Estimated); Study Completion 2024-05-18 (Estimated)

PRIMARY OUTCOMES:
PFS is determined by the IRC | 2 years
  Progression-free survival is determined by the IRC according to the RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No